CLINICAL TRIAL: NCT03505762
Title: A Randomized Phase II Pilot of Tailored Prednisone Reduction Versus Usual Care for the Treatment of Hyperglycemia During R-CHOP Chemotherapy
Brief Title: Tailored Prednisone Reduction in Preventing Hyperglycemia in Participants With B-Cell Non-Hodgkin Lymphoma Receiving Combination Chemotherapy Treatment
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00050108; NCI-2018-00585 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 98317 (Other: Wake Forest University Health Sciences); P30CA012197 (NIH)
Record Dates: First submitted 2018-04-12; First posted 2018-04-23 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Cyclophosphamide; Doxorubicin; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (tailored prednisone dose) (Experimental): Participants receive rituximab IV, vincristine sulfate IV, doxorubicin hydrochloride IV, and cyclophosphamide IV on day 1. Participants also receive tailored prednisone dose PO QD on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Prednisone; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Biological: Rituximab; Drug: Vincristine Sulfate
- Arm II (usual care prednisone dose) (Active Comparator): Participants receive rituximab, vincristine sulfate doxorubicin hydrochloride, and cyclophosphamide as in Arm I. Participants also receive usual care prednisone dose PO QD on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Prednisone; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
Other: Quality-of-Life Assessment — Ancillary correlative
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies how well tailored prednisone reduction works in preventing hyperglycemia in participants with B-cell non-Hodgkin lymphoma receiving combination chemotherapy treatment. Drugs used in chemotherapy, such as rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Reductions in prednisone dose may lower blood sugar levels.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the cumulative incidence of hyperglycemia after 3 cycles of treatment between standard or tailored rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate and prednisone (R-CHOP) chemotherapy.

SECONDARY OBJECTIVES:

I. To compare the cumulative incidence of hyperglycemia after 6 cycles of treatment and at 6 months post-treatment between standard or tailored R-CHOP chemotherapy.

II. To compare response rates after 6 cycles of treatment as measured by Cheson's criteria between standard or tailored R-CHOP chemotherapy.

III. To compare cumulative rates of grade III or higher adverse events using Common Terminology Criteria for Adverse Events (CTCAE) criteria between standard or tailored R-CHOP chemotherapy from cycle 1 through cycle 6.

IV. To compare severity of prednisone related adverse events using the Patient Reported Outcome (PRO)-CTCAE form between standard or tailored R-CHOP chemotherapy from cycle 1 through cycle 6.

V. To compare health related quality of life (HRQOL) between standard or tailored R-CHOP chemotherapy at baseline, cycle 4 day 1 and after cycle 6.

EXPLORATORY OBJECTIVES:

I. To evaluate the alternative glucose measures of fasting blood glucose (FBG), hemoglobin A1c (HbA1c), fasting insulin and fructosamine to estimate hyperglycemia.

II. To compare health related quality of life (HRQOL) in those with and without hyperglycemia after 3 cycles, 6 cycles, and 6 months post R-CHOP chemotherapy.

III. To compare glycemic variability between the standard and tailored prednisone arms at day 1 of each cycle IV. To determine the ability of patients in the standard or tailored prednisone R-CHOP groups to complete all six cycles of chemotherapy.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive rituximab intravenously (IV), vincristine sulfate IV, doxorubicin hydrochloride IV, and cyclophosphamide IV on day 1. Participants also receive tailored prednisone dose orally (PO) once daily (QD) on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Participants receive rituximab, vincristine sulfate doxorubicin hydrochloride, and cyclophosphamide as in Arm I. Participants also receive usual care prednisone dose PO QD on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of B cell non-Hodgkin lymphoma confirmed by World Health Organization (WHO) criteria
* Planned treatment with R-CHOP chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 3
* Life expectancy of greater than 3 months with chemotherapy
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document (either directly or via a legally authorized representative)

Exclusion Criteria:

* Uncontrolled human immunodeficiency virus (HIV), CD4 count < 50
* Diagnosis of primary central nervous system (CNS) lymphoma
* Unable to receive R-CHOP chemotherapy
* History of severe (i.e. anaphylactic) allergic reactions attributed to compounds of similar chemical or biologic composition to glucocorticoids and other component of R-
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection not controlled with antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia that cannot be rate controlled with medications, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with these agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of hyperglycemia of standard or tailored rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate and prednisone (R-CHOP) | After course 3 (63 days)
  Will use the Kaplan Meier method to estimate the cumulative incidence of hyperglycemia, and the log-rank test to compare hyperglycemia incidence by arm after 3 cycles of R-CHOP chemotherapy.

SECONDARY OUTCOMES:
Cumulative incidence of hyperglycemia of standard or tailored R-CHOP | Baseline up to 6 months
  Will use the Kaplan Meier method to estimate the cumulative incidence of hyperglycemia, and the log-rank test to compare hyperglycemia incidence by arm after 6 cycles and after 6 months of R-CHOP chemotherapy.
Response rates of standard or tailored R-CHOP as measured by Cheson's criteria | After of course 6 (126 days)
  Will use a Fisher's exact test to compare response rates after 6 cycles of R-CHOP by arm.
Rates of grade III or higher adverse events using Common Terminology Criteria for Adverse Events (CTCAE) criteria from standard or tailored R-CHOP | Up to 6 months
  Will compare the rates of the incidence of grade III and higher events by arm of R-CHOP for each cycle using Fisher's exact tests.
Severity of prednisone related adverse events using the Patient Reported Outcome (PRO)-CTCAE | Up to course 6 (126 days)
  Will compare the scoring of PRO-CTCAE assessments by arm of R-CHOP using two group t-tests at each time point of interest.
Health related quality of life (HRQOL) scores | Up to 6 months
  Evaluated using the Functional Assessment of Cancer Therapy (FACT)-Lymphoma, FACT Gynecologic Oncology Group-Neurotoxicity additional concerns and Patient-Reported Outcomes Measurement Information System 29. Will compare the HRQOL measures between arms receiving R-CHOP chemotherapy using two group t-tests at each time point of interest.

OTHER OUTCOMES:
Fasting blood glucose (FBG) levels | Up to 6 months
  Will examine glucose variability over time in FBG using linear mixed effects models to model between and with-person variation in glucose.
Hemoglobin A1C (HbA1c) levels | Up to 6 months
  Will examine glucose variability over time in HbA1c using linear mixed effects models to model between and with-person variation in glucose.
Fasting insulin | Up to 6 months
  Will examine glucose variability over time in fasting insulin using linear mixed effects models to model between and with-person variation in glucose.
Fructosamine levels | Up to 6 months
  Will examine glucose variability over time in fructosamine using linear mixed effects models to model between and with-person variation in glucose.
HRQOL scores in those with and without hyperglycemia | Up to 6 months
  Will compare quality of life between the those who are hyperglycemic and those that are not at cycle 3, cycle 6, and 12 months using a mixed model analysis covariance (ANCOVA) with adjustment for baseline quality of life.
Glycemic variability | Up to 6 months
  To compare glycemic variability between the arms, will model variability using mixed effect models of FBG and random blood glucose over time, allowing for differing within-person variance by arm as well as fitting a model with pooled variance and any characteristics that differ between the groups. Will use likelihood ratio tests to compare if there is greater variability in the tailored versus standard arms by comparing the pooled variance model to the model that allows the within-person variation to vary by arm.
Percentage of patients in the standard and tailored prednisone R-CHOP arms who complete all six cycles of chemotherapy | End of course 6 (126 days)
  Will compare the proportion of participants by arm using Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Rakhee Vaidya, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States